CLINICAL TRIAL: NCT02521909
Title: An in Vivo Evaluation of the ProMark, Root ZX II, and NRG Rider Electronic Apex Locators on the Accuracy of Working Length of Molars
Brief Title: Accuracy of Electronic Apex Locators ProMark, RootZX II and NRG Rider on Working Length of Multi-rooted Teeth
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Neville McDonald, Clinical Professor, Director of Endodontics, University of Michigan
Other Study IDs: HUM00093162
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Dental Pulp Diseases
Keywords: Root Canal length; Electronic apex locator; Endodontics
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Tooth Extraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tooth Extraction: Intervention is Tooth Extraction for Assessment of Different Apex Locators. All people in the study will contribute one or more teeth, which will be extracted for other clinical purposes, for device comparative testing
  Interventions: Device: ProMark (Tooth Extraction for Assessment of Different Apex Locators); Device: Root ZX II (Tooth Extraction for Assessment of Different Apex Locators); Device: NRG Rider (Tooth Extraction for Assessment of Different Apex Locators)

INTERVENTIONS:
Device: ProMark (Tooth Extraction for Assessment of Different Apex Locators) — The purpose of this study is to compare the accuracy of different apex locators on teeth that are scheduled for extractions. Before root canal therapy, dentists use a device called an electronic apex locator (EAL) to measure the root canal and to locate its opening at the tip of the tooth's root (called the apical foramen). A root canal is the space inside the root of a tooth. If the tissue within the root canal becomes infected, dentists may perform root canal therapy.
Device: Root ZX II (Tooth Extraction for Assessment of Different Apex Locators) — The purpose of this study is to compare the accuracy of different apex locators on teeth that are scheduled for extractions. Before root canal therapy, dentists use a device called an electronic apex locator (EAL) to measure the root canal and to locate its opening at the tip of the tooth's root (called the apical foramen). A root canal is the space inside the root of a tooth. If the tissue within the root canal becomes infected, dentists may perform root canal therapy.
Device: NRG Rider (Tooth Extraction for Assessment of Different Apex Locators) — The purpose of this study is to compare the accuracy of different apex locators on teeth that are scheduled for extractions. Before root canal therapy, dentists use a device called an electronic apex locator (EAL) to measure the root canal and to locate its opening at the tip of the tooth's root (called the apical foramen). A root canal is the space inside the root of a tooth. If the tissue within the root canal becomes infected, dentists may perform root canal therapy.

SUMMARY:
The purpose of this study is to compare the accuracy of different apex locators. Before root canal therapy, dentists use a device called an electronic apex locator (EAL) to measure the root canal and to locate its opening at the tip of the tooth's root (called the apical foramen). A root canal is the space inside the root of a tooth. If the tissue within the root canal becomes infected, dentists may perform root canal therapy.

DETAILED DESCRIPTION:
This study will generate data to compare the efficacy of three different manufactures of an instrument commonly used in dental clinics. The instruments are known as electronic apex locators (EAL). Electronic apex locators are used to measure the length of a root canal and to locate its opening at the end of the tooth's root (called the apical foramen). A root canal is the space inside the root of a tooth. If the tissue within the root canal becomes diseased, dentists may perform root canal therapy; for this reason the accuracy of the EAL is very important.

In this study patients who are scheduled for tooth extraction as part of their standard of care will be pre-screened by record review for candidacy as study subjects. If the scheduled patients screen as potentially eligible by reviewing their records, then they will be approached by the study team at the time of their pre-extraction consultation visit (this is a visit which occurs prior to the extraction visit). Only teeth scheduled to be extracted are suitable for this study. On the day of their standard of care tooth or teeth extraction(s) prior to the extraction the study team will conduct measurements with the EALs. After the EAL measurements the standard of care extractions will occur as standard of care, outside of the study, and by the patient's clinician. Extracted teeth will be given to the study team as long as they are not needed for further pathological review (extracted teeth are usually discarded and are rarely sent to a lab for further analysis). Also the teeth must be extracted without breaking. the study team will analyze them (ex-vivo) to generate true root measurements which will be compared to the data generated prior to extraction by the instruments which are the subject of this study. The instruments are the subject of this study, but in-vivo data generated by the instruments will be compared to ex-vivo data gained by measurements after the tooth/teeth is/are extracted.

ELIGIBILITY:
Inclusion criteria:

1. Be an adult over 18 years of age.
2. Multi-rooted teeth (molar or premolar) scheduled for extraction because of non-restorability, orthodontic or periodontal reasons
3. Be able to understand and provide informed consent for participation in the protocol

Exclusion criteria:

1. Any liver, kidney, heart, blood, metabolic or systemic disease which may make execution of the protocol or interpretation of the results difficult
2. History of syphilis, HIV, Hepatitis B or Hepatitis C
3. Pregnant
4. Currently receiving radiation
5. Any other medical/physical condition the PI deems unacceptable for participation.
6. Patient unable to provide informed consent
7. Plan to participate in another clinical trial within 30 days of entrance into this study
8. Tooth with "non-intact crown"
9. Presence of an electronic implantable device (pacemaker, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals in need of extraction of multi-rooted teeth
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Tooth Length Measurement after extraction | 48 hours After Extraction
  A Kodak 9000 3D is used as a small-volume field of view (FOV) CBCT based on its scan to allow cone beam reconstructions at 0.076 mm with a minimal discrepancy compared to histologic sections. The extracted teeth are imaged and slices reviewed for accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Neville McDonald, BDS, MS, Principal Investigator — University of Michigan
Locations (1):
- U of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No